CLINICAL TRIAL: NCT05661110
Title: Integrated Biomarker Analysis for Hyperthermic Intraperitoneal Chemotherapy(HIPEC) Combined PD1/PDL1 Inhibitor Treatment in Patients of Advanced Gastric Cancer With Peritoneal Metastasis
Brief Title: Biomarker Analysis of HIPEC Combined With PD1/PDL1 Inhibitor for Gastric Cancer With Peritoneal Metastasis
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: HIPEC-11
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer
Keywords: Biomarker
MeSH Terms: conditions — Stomach Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and residual tissue from surgery or tumor biopsy will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Sample Collection: Prospective sample collection from participants treated with HIPEC combined PD1/PDL1inhibitor at Affiliated Cancer Hospital & Institute of Guangzhou Medical University under standard of care treatment. Blood and tissue samples will be collected prior to initiation of conversion therapy. And thereafter at the four time points: before and after surgery(±7 days), before the start of the second cycle of adjuvant, tumour progression, blood sample will be collected too.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — All patients will be treated with standard of conversion treatment with HIPEC combined PD1/PDL1 inhibitor. After obtaining written informed consent, participants will have serial blood, tumor tissue collection. The blood collection (10 ml) should coincide with routine clinical blood draw to minimize participant discomfort if possible. No additional procedures will be performed other than phlebotomy. Participants will remain on the study for as long as they are being followed or treated at Affiliated Cancer Hospital & Institute of Guangzhou Medical University. Participants can withdraw from the study at any time.

SUMMARY:
A single-center, observational study, integrated biomarker analysis of HIPEC combined Programmed cell death 1 /Programmed cell death 1 ligand 1(PD1/PDL1)inhibitor in previously treated patients of advanced gastric cancer with peritoneal metastasis. Tests will be performed on tumor tissue and blood samples, and imaging assessments will be reviewed in order to monitor how well each patient responds to treatment. This is an observational study, so participants will not receive cancer treatment, other than the treatment received as standard of care.

DETAILED DESCRIPTION:
To analyze the correlation between genomic alterations, gene expression characteristics and the efficacy of HIPEC combined with PD1/PDL1 inhibitor conversion therapy in patients with peritoneal metastasis of gastric cancer. Circulating tumor DNA(ctDNA) in plasma samples and DNA, RNA in tumor tissue sample were obtained over the course of HIPEC combined PD1/PDL1 inhibitor conversion treatment will be assessed by high-intensity, next-generation sequencing(NGS) to identify genomic alterations. The assay will performed used AmoyDx® Master Panel(Amoy Diagnostics Co., Xiamen, China), which contains 559 genes for DNA mutation detection and 1813 genes for RNA expression and fusion detection. Data acquired will be analyzed to characterize the association between these genetic elements, clinical response, and durability of responses. There will be prospective groups for the study. Samples will be collected from patients in the prospective cohort who have been treated with HIPEC combined PD1/PDL1 inhibitor at Affiliated Cancer Hospital & Institute of Guangzhou Medical University under standard of conversion treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced gastric (gastroesophageal junction) adenocarcinoma confirmed by histology;
2. Age 18-75 years, Male or Non-pregnant female
3. Eastern Cooperative Oncology Group(ECOG): 0~1；
4. Negative for human epidermal growth factor receptor 2(HER-2) by immunocytochemistry or fluorescence in situ hybridization；
5. The presence of gastric cancer peritoneal metastasis is confirmed by laparoscopic exploration, and the PCI≤20；
6. Patients had received HIPEC combined with PD1/PDL1 inhibitor conversion therapy.
7. Signed the Informed Consent Form, and blood and tissue samples can be obtained;

Exclusion Criteria:

1. Other distal metastases besides peritoneal metastases (e.g., liver, lung, pleural, brain, bone metastases, etc.);
2. Other patients who were considered unsuitable for inclusion by the researchers;

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Advanced gastric adenocarcinoma confirmed by histology with peritoneal metastasis
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between the status, numerical changes of ctDNA during HIPEC combined with PD1/PDL1 inhibitor conversion therapy and postoperative R0 resection rate. | 3 months
  R0 resection rate refers to the proportion of all patients with negative margins under the microscope of tumor specimens after surgery to the total number of participants. To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during treatment.

SECONDARY OUTCOMES:
Genomic changes of ctDNA and see if they are predictive of ORR. | 3 months
  Objective response rate(ORR): ORR = (number of subjects with complete response (CR) + partial response (PR))/total number of subjects ×100%. Measurable lesion according to the Response Evaluation Criteria In Solid Tumours(RECISTv1.1). To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during treatment.
Genomic changes of ctDNA and see if they are predictive of overall survival time. | 2 years
  Overall survival time(OS) refers to the time of first use of the drug to the time of death. At the end of the study, if the subject is still alive, refer the known "date of last survival of the subject" as the date of censoring. To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during and after treatment.
Genomic changes of ctDNA and see if they are predictive of event-Free Survival. | 2 years
  Event-Free Survival(EFS): Defined as the interval between the first conversion therapy and the first recorded related events, including preoperative disease progression, postoperative disease recurrence, and death from any cause. To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during and after treatment.
Genomic changes of ctDNA and see if they are predictive of relapse-Free Survival. | 2 years
  Relapse-Free Survival(RFS): Defined as postoperative the first recorded postoperative recurrence of disease or death from any cause. To dynamically evaluate the ctDNA profiles by next-generation sequencing and illustrate the genomic changes of ctDNA at baseline, during and after treatment.

OTHER OUTCOMES:
Genetic and transcriptional profiling results. | From baseline (prior to initiation of conversion therapy)
  Mutation and transcriptomic information will be recorded by NGS using AmoyDx® Master Panel, which contains 559 genes for DNA mutation detection and 1813 genes for RNA expression and fusion detection.

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, Doctor, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leal A, van Grieken NCT, Palsgrove DN, Phallen J, Medina JE, Hruban C, Broeckaert MAM, Anagnostou V, Adleff V, Bruhm DC, Canzoniero JV, Fiksel J, Nordsmark M, Warmerdam FARM, Verheul HMW, van Spronsen DJ, Beerepoot LV, Geenen MM, Portielje JEA, Jansen EPM, van Sandick J, Meershoek-Klein Kranenbarg E, van Laarhoven HWM, van der Peet DL, van de Velde CJH, Verheij M, Fijneman R, Scharpf RB, Meijer GA, Cats A, Velculescu VE. White blood cell and cell-free DNA analyses for detection of residual disease in gastric cancer. Nat Commun. 2020 Jan 27;11(1):525. doi: 10.1038/s41467-020-14310-3. PMID 31988276
- [Background] Wang D, Cabalag CS, Clemons NJ, DuBois RN. Cyclooxygenases and Prostaglandins in Tumor Immunology and Microenvironment of Gastrointestinal Cancer. Gastroenterology. 2021 Dec;161(6):1813-1829. doi: 10.1053/j.gastro.2021.09.059. Epub 2021 Oct 2. PMID 34606846
- [Background] Smyth EC, Gambardella V, Cervantes A, Fleitas T. Checkpoint inhibitors for gastroesophageal cancers: dissecting heterogeneity to better understand their role in first-line and adjuvant therapy. Ann Oncol. 2021 May;32(5):590-599. doi: 10.1016/j.annonc.2021.02.004. Epub 2021 Feb 17. PMID 33609722